CLINICAL TRIAL: NCT00449579
Title: The Diagnostic Benefits of the HyperQTM System in ECG Stress Testing
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Collaborators: BSP Biological Signal Processing Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MAC_01
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2006-10

CONDITIONS: Myocardial Ischemia
Keywords: Ischemia; Myocardial; HF-ECG
MeSH Terms: conditions — Myocardial Ischemia; Ischemia

INTERVENTIONS:
Device: Excercise stress test with high frequency ECG recording (HyperQ™ System)

SUMMARY:
The main objective of this study is to determine the usefulness of the HyperQ™ System in improving the positive predictive value of conventional ECG stress testing.

Patients who are referred for stress test will perform an ECG stress test on a treadmill, with high-frequency ECG recording from conventional 12 leads using BSP's HyperQ™ System. Conventional 12 lead ECG, as well as HyperQ™ recordings will be provided by the HyperQ™ System. The results of the conventional test and the HyperQ™ data will be compared, using one of three cardiac tests (stress echocardiography, SPECT myocardial perfusion imaging and angiography) as gold standards.

Statistical analysis will compare the sensitivity, specificity, PPV and NPV of the conventional and HyperQ™ stress ECG in detecting myocardial ischemia.

DETAILED DESCRIPTION:
The study population will comprise of 1200 patients referred to stress test in three Maccabi clinics or cardiac medical centers. All patients will perform an ECG stress test with high-frequency ECG recording from conventional 12 leads using BSP's HyperQ™ System. The recording will be done without affecting or interfering with any aspect of the normal due course of the test. Standard Bruce protocol or modified Bruce protocol will be used, with standard test termination indications. Two minutes of rest ECG will be recorded prior to stating the protocol.

Following the test, the physician will interpret the test's results in the conventional manner (e.g. ST changes, chest pain, etc) and decide whether the subject should be referred to additional tests.

HyperQ™ data will be analyzed in two phases: (i) Interpretation by the physician in a non-blinded manner one day following the stress test and (ii) after performing all the exercise tests of the study group, blindly to the conventional diagnosis and the HyperQ™ analysis done previously, as well as to other outcomes of imaging procedures. The first HyperQ™ reading will be used to detect the subjects who were positive according to the HyperQ™ system but negative according to the conventional stress testing. These subjects will be referred by the physician to further clinical investigation. The first reading will also be used to assess the physician's interpretation in a scenario that represents a realistic clinical setting, while the second reading will be used to examine the unbiased clinical benefit of HyperQ™ data.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred to stress ECG
* Subjects age ≥ 45
* Subject signed an Informed Consent form

Exclusion Criteria:

* Subject with contraindications for stress ECG
* Subject with implantable pacemaker or defibrillator
* Subject with LBBB
* Subject with QRS duration ≥ 110 mSec
* Subject with Wolff-Parkinson-White Syndrome

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2006-08; Study Completion 2007-10

PRIMARY OUTCOMES:
ST changes
HyperQ results

CONTACTS AND LOCATIONS:
Overall Officials: Haim Silber, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Dr. Silber Clinic, Kfar Saba, Israel

REFERENCES:
- See also: HyperQ Technology by BSP Ltd. — http://www.bsp.co.il